CLINICAL TRIAL: NCT02301130
Title: Phase 1 Study of Mogamulizumab (KW-0761) in Combination With MEDI4736 (Durvalumab) and Mogamulizumab in Combination With Tremelimumab in Subjects With Advanced Solid Tumors
Brief Title: Study of Mogamulizumab + MEDI4736 (Durvalumab) and Mogamulizumab + Tremelimumab in Subjects w/ Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0761-012
Record Dates: First submitted 2014-11-21; First posted 2014-11-25 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors
Keywords: advanced solid tumors; solid tumors; mogamulizumab; MEDI4736 (Durvalumab); Tremelimumab; POTELIGEO®; KW-0761
MeSH Terms: interventions — mogamulizumab; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mogamulizumab + MEDI4736 (Durvalumab) (Experimental): During Parts 1 and 2, mogamulizumab and MEDI4736 (Durvalumab) are administered at appropriate intervals.
  Part 1 (Dose Escalation Phase)
  - During Cohort 1A to 4A, increased doses of mogamulizumab and MEDI4736 (Durvalumab) are administered.
  Part 2 (Cohort Expansion Phase)
  * Patients will be treated with maximum tolerated dose established in the Dose Escalation Phase for each combination.
  Interventions: Biological: mogamulizumab; Biological: MEDI4736 (Durvalumab)
- mogamulizumab + tremelimumab (Experimental): During Parts 1 and 2, mogamulizumab and tremelimumab are administered at appropriate intervals.
  Part 1 (Dose Escalation Phase)
  - During Cohort 1B to 4B, increased doses of mogamulizumab and tremelimumab are administered.
  Part 2 (Cohort Expansion Phase)
  * Patients will be treated with maximum tolerated dose established in the Dose Escalation Phase for each combination.
  Interventions: Biological: mogamulizumab; Biological: tremelimumab

INTERVENTIONS:
Biological: mogamulizumab — Mogamulizumab will be administered intravenously (IV).
  Other Names: KW-0761; POTELIGEO®
Biological: MEDI4736 (Durvalumab) — MEDI4736 will be administered intravenously (IV).
  Other Names: Durvalumab
  Arms: mogamulizumab + MEDI4736 (Durvalumab)
Biological: tremelimumab — Tremelimumab will be administered intravenously (IV).
  Other Names: ticilimumab; CP-675,206
  Arms: mogamulizumab + tremelimumab

SUMMARY:
Mogamulizumab in Combination with MEDI4736 (Durvalumab) and Mogamulizumab in Combination with Tremelimumab in Subjects with Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Locally advanced or metastatic solid tumors;
* Histologically or cytologically confirmed disease;
* Failed or were intolerant to at least one prior systemic treatment regimen with oral or IV medications and have no additional therapy options known to prolong survival with the exception of PD-1 or PD-L1 blockade therapy for subjects who will be enrolled in treatment arm A. Subjects with non-small cell lung cancer must have received at least one platinum doublet regimen. Subjects with known epidermal growth factor receptor tyrosine kinase inhibitor activating mutations or anaplastic lymphoma kinase rearrangement must have also exhausted approved targeted therapy options;
* The subject has a tumor suitable for biopsy and is willing to undergo tumor biopsy, preferably of the primary tumor, within 28 days prior to Cycle 1/Visit Day 1;

Exclusion Criteria:

* Any concurrent chemotherapy, biologic, hormonal, radiation, or investigative therapy for cancer treatment within 21 days prior prior or within 6 weeks prior to Cycle 1/Visit Day 1 for nitrosoureas or mitomycin C;
* Concurrent or prior use of immunosuppressive medication within 28 days;
* Active or prior documented autoimmune, or inflammatory bowel disease, or inflammatory bowel disease. or systemic treatment for psoriasis within the past 5 years.;
* Prior hypersensitivity reaction to monoclonal antibodies, other therapeutic proteins, or immunotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11-26 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting adverse events | Screening through 90 days after the last dose of study medication
Number of subjects reporting serious adverse events | Screening through 90 days after the last dose of study medication
Percentage of subjects reporting serious adverse events | Screening through 90 days after the last dose of study medication
Percentage of subjects reporting adverse events | Screening through 90 days after the last dose of study medication
Number of subjects experiencing dose-limiting toxicity | First dose of study medications through 4 weeks after the last dose of study medication

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - The Angeles Clinic, Los Angeles, California
  - UCLA Hematology & Oncology Clinic, Los Angeles, California
  - Yale Cancer Center, New Haven, Connecticut
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Georgia Cancer Center, Augusta, Georgia
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Zamarin D, Hamid O, Nayak-Kapoor A, Sahebjam S, Sznol M, Collaku A, Fox FE, Marshall MA, Hong DS. Mogamulizumab in Combination with Durvalumab or Tremelimumab in Patients with Advanced Solid Tumors: A Phase I Study. Clin Cancer Res. 2020 Sep 1;26(17):4531-4541. doi: 10.1158/1078-0432.CCR-20-0328. Epub 2020 Jun 25. PMID 32586937